CLINICAL TRIAL: NCT01529879
Title: A Prospective Randomized-Controlled Evaluation of an Implant System With a Novel Abutment Attachment Design for the Preservation of Crestal Bone
Brief Title: Assessment of the Effect of an Implant System With a Novel Abutment Attachment Design on Crestal Bone Preservation
Acronym: Polaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3014
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: edentulism; dental implants; clinical study; Nanotite Certain Tapered implant; randomized; crestal bone level
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New abutment connection implant (Experimental): Implant with new abutment connection
  Interventions: Device: New Abutment Connection implant
- Nanotite Certain Tapered implant (Active Comparator): Nanotite Certain Tapered (standard abutment connection) implant
  Interventions: Device: Nanotite Certain Tapered implant

INTERVENTIONS:
Device: New Abutment Connection implant — New abutment connection implant
  Other Names: Osseotite Endosseous dental implant
  Arms: New abutment connection implant
Device: Nanotite Certain Tapered implant — Nanotite Certain Tapered (standard abutment connection) implant
  Other Names: Nanotite endosseous dental implant
  Arms: Nanotite Certain Tapered implant

SUMMARY:
Integration success rates and the preservation of crestal bone will be higher for the experimental device than for the control implants.

DETAILED DESCRIPTION:
In this study patients are randomized to receive either the experimental implant system or the control Nanotite Certain Tapered (standard abutment connection) and assessed for integration success measured by lack of implant mobility and lack of bone loss obtained at various study time points

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and older than 18 years of age
* patients needing at least one dental implant to treat partial edentulism
* patients physically able to tolerate surgical and restorative dental procedures
* patients agreeing to all protocol visits

Exclusion Criteria:

* patients with infection or severe inflammation at the intended treatment sites
* patients smoking greater than 10 cigarettes per day
* patients with uncontrolled diabetes mellitus
* patients with uncontrolled metabolic diseases
* patients who received radiation treatment to the head in the past 12 months
* patients needing bone grafting at the intended treatment sites
* patients known to be pregnant at screening visit
* patients with para-functional habits like bruxing and clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cumulative success rate | 2 years
  Crestal bone regression (amount of bone loss measured) and equivalence in integration success (implant mobility)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Arango, DDS, Principal Investigator — Institucion Universitaria Colegios de Colombia
Locations (1):
- UNICOC, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No